CLINICAL TRIAL: NCT00666250
Title: Effects of Xoçai Antioxidant Supplements on Atherosclerosis Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Xocai01
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension; Dyslipidemia; Hyperglycemia
Keywords: blood pressure; dyslipidemia; hyperglycemia
MeSH Terms: conditions — Hypertension; Dyslipidemias; Hyperglycemia | interventions — Chocolate; whole grape extract; blueberry extract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline (No Intervention): Baseline values off chocolate supplement
- Low Dose (Experimental): Low dose of dietary supplement 30 ml tid (Activ Xocai Drink)
  Interventions: Dietary Supplement: Xocai Activ drink
- High-dose (Experimental): High dose of dietary supplement 90 ml tid (Xocai Activ drink)
  Interventions: Dietary Supplement: Xocai Activ drink

INTERVENTIONS:
Dietary Supplement: Xocai Activ drink — proprietary blend of cocoa powder and extracts of acai, grape and blueberry
  Other Names: Xocai Activ drink;; cocoa powder,; acai extract,; grape extract,; blueberry extract
  Arms: High-dose; Low Dose

SUMMARY:
An antioxidant dietary supplement made from cocoa powder, and extracts of acai, grape and blueberry will be tested for effects on blood sugar, blood pressure, cholesterol and related parameters in human subjects.

DETAILED DESCRIPTION:
Background and Introduction It has long been known that increased intake of plant products results in reduced risk of atherosclerosis and cardiovascular disease, which are the most important causes of death and disability in Western societies. This protective effect has been found to correlate with increased plasma levels of various antioxidant vitamins along with the expected increased resistance of the plasma to oxidation, and reduced evidence of oxidation of lipoproteins and other plasma components. It also has long been understood that oxidized LDL, and related lipoproteins which also contain apo B-100, are a primary driving force in the process of atherogenesis. These two facts have led to a very strong interest in developing antioxidant treatments as likely effective atheropreventive measures. This quest has taken the form of several large, long-term interventional studies, in which patients have been given purified antioxidant vitamins in an effort to reduce cardiovascular events. Surprisingly, almost without exception these interventions have failed to show any favorable effects. The cause of this paradox remains unknown, but may have resulted either from the reliance on antioxidant vitamins, rather than other antioxidant elements in the diet, or from the use of highly purified products, instead of more lightly processed food elements.

Cocoa mass (or cocoa powder in the dried form) is the edible non-fat part of the cacao bean which remains once the fatty cocoa butter has been removed. Cocoa mass or powder is a rich source of polyphenol antioxidants of the flavonoid family. The predominant flavonoids in cocoa are flavonols, including both the oligomeric proanthocyanidins (procyanidins and prodelphinidins) and the monomeric catechins and epicatechins. Recent studies have shown that chocolate preparations which are high in cocoa (and thus high in flavonol content) may have several beneficial effects on the vasculature and on various risk factors for atherosclerosis. These likely beneficial effects include:

1. Increased vascular reactivity
2. Improved arterial compliance
3. Increased HDL-C levels,
4. Decreased oxidation of LDL, and
5. Reduced insulin resistance.

Although several of these studies have compared preparations with low vs. high content of cocoa (or flavonols), only one study of which we are aware has tested effects of a source of chocolate other than a high-fat chocolate bar. Only a non-bar product can readily exclude cocoa butter and/or butterfat and thus be low in fat content. Meanwhile the relatively high fat content of a chocolate bar, even if made with high cocoa powder content (thus a "dark" chocolate bar) adds many calories to the product and may well reduce the beneficial effects of the cocoa. Apparently also, all of the preparations tested in the published studies were relatively high in sugar content, which also adds calories and may reduce the benefits of the cocoa.

In addition there are many inconsistencies among studies of standard chocolate preparations regarding the above-mentioned beneficial effects (for example, studies failing to show lipid or anti-inflammatory effects), and these inconsistencies may relate to various issues. First, of all the elements in chocolate-containing foods, cocoa mass or powder appears to contain virtually all of the antioxidant factors. Variability in cocoa powder content, or possible blunting of its benefits by the addition of variable amounts of cocoa butter might variably reduce the beneficial effects. Second, the alkaline processing of cocoa (which is routine for virtually all bar and powdered chocolate products) may reduce its antioxidant content and activity. Thus, the variability in published results among various chocolate preparations could be due to differences in the degree and type of processing of the cocoa (and resulting differences in its antioxidant content), and/or differences in the presence of other components (such as fat and/or sugar) which might block beneficial effects of the cocoa.

Açai fruit appears to have even greater content of antioxidant polyphenols (primarily as anthocyanins) than does cocoa mass or powder, especially when preserved from fresh açai juice as freeze-dried açai powder. Açai is known to contain many vitamins and minerals as well as some fats, and is a rich source of phytosterols. It is said to be able to lower LDL levels, likely because of its unsaturated and monounsaturated fat content. It is also said to have anti-inflammatory effects. Although processing into freeze-dried açai powder removes most of the fat, phytosterols and dietary fiber, the unique potential of açai appears to be primarily in its many anthocyanin antioxidants, which are best preserved in the freeze-dried powder. Unfortunately, in contrast to the many studies on chocolate, there appear to be no published scientific studies of physiologic effects of Açai (as an antioxidant or otherwise) in humans. A recent lay review of açai by Alexander G. Schauss, PhD, FACN ("Açai: The Nutritional and Antioxidant-Rich Amazonian Palm Tree Fruit," Sound Concepts, 2005), states that some human studies have been performed with açai and that the first scientific articles are currently in preparation. Dr Schauss does not mention, however, any detail about the methods or results of any such studies.

Blueberries, grapes and peppers have natural antioxidants, albeit in far lesser quantities than acai. With the exception of grapes, the in vivo effects of these antioxidant-rich fruits on human subjects have been very little studied. Research into the intake of alcoholic and non-alcoholic grape products (both from lighter- and darker-colored grapes) has shown significant antioxidant effects, especially with dark grapes. Any effects of grapes on atherosclerosis or its many standard risk factors remain controversial at best, and in many cases are unknown. Given the encouraging scientific data regarding antioxidant and vascular effects of cocoa and grapes in human subjects, further studies of non-vitamin antioxidant-rich food products are clearly warranted.

The study product, Xoçai Activ drink , has been carefully designed to try to maximize antioxidant content and effects in a pleasant-tasting natural food product. It achieves this by (1) including many ingredients with naturally high antioxidant content, cocoa powder, and Acai, grape and blueberry powders. (2) minimizing the processing of its components, and (3) eliminating added fat both to minimize potential interference with the likely favorable effects of its main ingredients, and to minimize its total caloric content.

In light of the high antioxidant content (manifested as high ORAC, etc.) of Xoçai Activ it is a prime candidate for studies of antioxidant effects in humans in vivo. If this study can show significant effects on clinical-relevant endpoints, such as lipids, glucose tolerance, blood pressure, or vascular function, it would indicate that clinical disease can be prevented with antioxidant supplement therapy.

Objectives:

Hypotheses

We hypothesize that when given to human subjects:

1. Xoçai Activ will have dose-dependent antioxidant effects in human subjects
2. Xoçai Activ will improve several atherosclerosis risk factors in a dose-dependent manner:

Specific Aims We will perform an open-label pilot dose-response study which we will test our hypotheses by measuring various individual factors related to the above aims.

All of the study parameters will be measured at baseline and at the end of two treatment periods of two weeks each, one at low dose (1 square three times/d) and high dose (two squares three times/d). The study will last about 5 weeks, counting the screening portion.

Patient Selection Criteria Subjects for the study will be up to 5 men and 5 women. All subjects will be from 18-79 years of age, with a body mass index <35, and of good general health. Subjects will be excluded if they regularly use lipid-altering medications (including niacin over 100 mg/d and DHA/EPA over one gram/d), alcohol, tobacco or antioxidant supplements (other than a standard multiple vitamin) and if they have a history of active liver, renal, or thyroid disease, or active cancer.

Study Design:

The study will be done with up to 10 subjects with endpoints measured at screening, baseline and then every 2 weeks for 4 weeks of treatment. The first two weeks of the study, participants will be instructed to drink three one-ounce servings of Xocai Activ a day. The second two weeks, participants will be instructed to drink three three-ounce servings of Xocai Activ a day (nine ounces daily). Subjects will be carefully instructed how to mix the dry Xocai Activ powder with the correct amount of water so that the proper amount of Xocai Activ will be consumed during both the low- and high-dose periods. There will be a total of 7 clinic visits with a total of 470 mL of blood taken.

Due to the difficulty in preparing placebo interventions, this study will not be double-blinded. We will however, blind the measurement of all laboratory assays.

Study Endpoints:

All blood and urine will be taken, and all vascular and body composition measurements will be performed after a 12-hour overnight fast twice during the baseline period and twice at the end of each 2-week period of intervention.

Diet: Subjects will have their routine diet assessed between the two baseline visits, and at the end of the study by means of a 3-day food record. They will be instructed to consume no antioxidant supplements, and to minimize consumption of high antioxidant foods (chocolate, blueberries, red grapes, etc.) during the study.

Laboratory measurements: Antioxidant levels and activity are a primary endpoint of the study and will be measured at baseline and in each dose in each subject.

Vascular measurements: Blood pressure and vascular function should be favorably affected by Xoçai, and they will be measured by standard, established methods in our research clinic.

Body composition: We anticipate that the effects of Xoçai may be determined in part by body composition, in that more obese subjects, who have greater abnormalities in oxidation, inflammation, lipids and vascular function, will have a greater response. We will measure body composition by percent body fat by bioelectrical impedance.

Study data will be obtained in the laboratory by Dr. Nanjee and will be analyzed by all investigators. Confidentiality will be maintained by not divulging personal information beyond those directly involved in subject contact and data collection, and by maintaining hard copies of subject records in locked files. Computer files with personal information identifying subjects will be kept exclusively in secure password-protected computer files. Data analysis will be performed using files identifying patients only by subject number.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult not taking cocoa supplements

Exclusion Criteria:

* diabetes mellitus

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 weeks

SECONDARY OUTCOMES:
Plasma Lipids | 4 weeks
Arterial Compliance | 4 weeks
Fasting and post-challenge glucose and insulin | 4 weeks
urine microalbumin/creatinine ratio | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eliot Brinton, MD, Principal Investigator — University of Utah
Locations (1):
- Cardiovascular Genetics, University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- See also: Cardiovascular Genetics, University of Utah — http://utah.edu